CLINICAL TRIAL: NCT05552222
Title: A Phase 3 Randomized Study Comparing Teclistamab in Combination With Daratumumab SC and Lenalidomide (Tec-DR) and Talquetamab in Combination With Daratumumab SC and Lenalidomide (Tal-DR) Versus Daratumumab SC, Lenalidomide, and Dexamethasone (DRd) in Participants With Newly Diagnosed Multiple Myeloma Who Are Either Ineligible or Not Intended for Autologous Stem Cell Transplant as Initial Therapy
Brief Title: A Study of Teclistamab in Combination With Daratumumab and Lenalidomide (Tec-DR) and Talquetamab in Combination With Daratumumab and Lenalidomide (Tal-DR) in Participants With Newly Diagnosed Multiple Myeloma
Acronym: MajesTEC-7
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109237; 64007957MMY3005 (Other: Janssen Research & Development, LLC); 2022-000909-28 (EudraCT Number); 2023-503442-30-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05463939 (Approved for marketing)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone; talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Teclistamab, Daratumumab SC, and Lenalidomide (Tec-DR) (Experimental): Participants will receive teclistamab as subcutaneous (SC) injection in combination with daratumumab and lenalidomide.
  Interventions: Drug: Teclistamab; Drug: Daratumumab; Drug: Lenalidomide
- Talquetamab, Daratumumab SC, and Lenalidomide (Tal-DR) (Experimental): Participants will receive talquetamab as SC injection in combination with daratumumab and lenalidomide.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Talquetamab
- Daratumumab SC, Lenalidomide, and Dexamethasone (DRd) (Active Comparator): Participants will receive daratumumab as SC injection with lenalidomide and dexamethasone.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered as SC injection.
  Other Names: JNJ-64007957
  Arms: Teclistamab, Daratumumab SC, and Lenalidomide (Tec-DR)
Drug: Daratumumab — Daratumumab will be administered as SC injection.
Drug: Lenalidomide — Lenalidomide will be administered orally.
Drug: Dexamethasone — Dexamethasone will be administered either orally or intravenously (IV).
  Arms: Daratumumab SC, Lenalidomide, and Dexamethasone (DRd)
Drug: Talquetamab — Talquetamab will be administered as SC injection.
  Other Names: JNJ-64407564
  Arms: Talquetamab, Daratumumab SC, and Lenalidomide (Tal-DR)

SUMMARY:
The purpose of this study is to compare the efficacy of teclistamab in combination with daratumumab and lenalidomide (Tec-DR) and talquetamab in combination with daratumumab and lenalidomide (Tal-DR) versus daratumumab, lenalidomide, dexamethasone (DRd).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of multiple myeloma according to the International Myeloma Working Group (IMWG) diagnostic criteria
* Be newly diagnosed and not considered a candidate for high-dose chemotherapy with autologous stem cell transplant (ASCT) due to: ineligible due to advanced age OR; ineligible due to the presence of comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with ASCT OR; deferral of high-dose chemotherapy with ASCT as initial treatment
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
* A participant must agree not to be pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment
* A participant must agree not to plan to father a child while enrolled in this study or within 100 days after the last dose of study treatment

Exclusion Criteria:

* Received any prior therapy for multiple myeloma or smoldering myeloma other than a short course of corticosteroids (not to exceed total of 160 milligrams [mg] dexamethasone or equivalent). In addition, received a cumulative dose of systemic corticosteroids equivalent to greater than or equals to (>=) 20 mg of dexamethasone within 14 days before randomization
* Had plasmapheresis within 28 days of randomization
* Had a stroke, transient ischemic attack, or seizure within 6 months prior to randomization
* Known allergies, hypersensitivity, or intolerance to teclistamab or talquetamab excipients
* Known contraindications to the use of daratumumab or lenalidomide per local prescribing information
* Myeloma Frailty Index of >=2 with the exception of participants who have a score of 2 based on age alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2031-04-30 (Estimated); Study Completion 2033-10-28 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From randomization to the date of disease progression or death (Up to 09 years)
  PFS is defined as the duration from the date of randomization to either progressive disease or death, whichever comes first. Disease progression will be determined according to the International Myeloma Working Group (IMWG) response criteria.
12-Month Minimal Residual Disease (MRD)-Negative Complete Response (CR) | At Month 12
  12-month MRD-negative CR is defined as participants who achieve MRD-negative status at 12 months, as determined by next-generation sequencing (NGS) with sensitivity of 10^-5, prior to progressive disease or subsequent anti-myeloma therapy and who also achieve CR or better, according to IMWG criteria.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better | From randomization up to 09 years
  VGPR or better is defined as the percentage of participants achieving VGPR and CR (including stringent complete response [sCR]) prior to subsequent antimyeloma therapy in accordance with the IMWG criteria during or after the study treatment.
Complete Response (CR) or Better | From randomization up to 09 years
  CR or better is defined as the percentage of participants achieving CR or sCR prior to subsequent antimyeloma therapy in accordance with the IMWG criteria during or after the study treatment.
Sustained Minimal Residual disease (MRD)-negative Complete Response (CR) | From randomization up to 09 years
  Sustained MRD-negative CR is defined as participants with CR or better who sustain MRD-negative status, as determined by NGS with sensitivity of 10^-5, for at least 12 months without any examination showing MRD positive status or progressive disease in between.
MRD-negative CR | From randomization up to 09 years
  MRD-negative CR is defined as the percentage of participants who achieve MRD-negative status, as determined by NGS with sensitivity of 10^-5, at any time after randomization and prior to progressive disease or subsequent antimyeloma therapy and who achieve CR or better.
Progression Free Survival on Next-line Therapy (PFS2) | From randomization up to 09 years
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as progressive disease as assessed by investigator that starts after the next line of subsequent therapy, or death from any cause, whichever occurs first.
Overall Survival (OS) | From randomization to the date of death (up to 09 years)
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Number of Participants with Adverse Events (AEs) by Severity | From randomization up to 09 years
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening, and Grade 5: death related to adverse event.
Number of Participants with Abnormalities in Laboratory Parameters | From randomization up to 09 years
  Number of participants with abnormalities in laboratory parameters (serum chemistry and hematology) will be reported.
Number of Participants with Abnormalities in Vital Signs | From randomization up to 09 years
  Number of participants with abnormalities in vital signs (temperature, pulse/heart rate, respiratory rate, blood pressure) will be reported.
Number of Participants with Abnormalities in Physical Examination | From randomization up to 09 years
  Number of participants with abnormalities in physical examination will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | From randomization up to 09 years
  Number of participants with abnormalities in ECG will be reported.
Serum Concentrations of Teclistamab and Talquetamab | From randomization up to 09 years
  Serum samples will be analyzed to determine concentrations of teclistamab and talquetamab using validated, specific, and sensitive methods.
Number of Participants with Anti-drug Antibodies (ADAs) to Teclistamab and Talquetamab | From randomization up to 09 years
  Number of participants with ADAs to teclistamab and talquetamab will be reported.
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) | From baseline up to 9 years
  The EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from Baseline in Treatment-related Symptoms as Assessed by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline through Cycle 6 (each cycle of 28 days) (up to 196 days)
  The National Cancer Institute's (NCI's) PRO-CTCAE is an item library of common AEs experienced by people with cancer that are appropriate for self-reporting of treatment tolerability. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference of the AEs. It ranges from 0 to 4 with higher scores indicating higher frequency or greater severity/impact.
Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | From baseline up to 9 years
  The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time to Sustained Worsening in Symptoms, Functioning, and HRQoL | From randomization up to 09 years
  Time to sustained worsening in symptoms, functioning and HRQoL is defined as the interval from the date of randomization to the start date of meaningful change.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (257):
- United States (55):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCSF Fresno, Clovis, California
  - City of Hope Cancer Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of Connecticut, Farmington, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - ChristianaCare Helen F Graham Cancer Center and Research Institute, Newark, Delaware
  - Cleveland Clinic Florida, Weston, Florida
  - City of Hope Cancer Center, Newnan, Georgia
  - University Of Illinois Medical Center, Chicago, Illinois
  - University of Iowa Health Care, Waukee, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - LSUHSC Shreveport Feist-Weiller Cancer Center, Shreveport, Louisiana
  - Johns Hopkins University School of Medicine JHUSOM, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Cancer - Detroit Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Cancer And Hematology Centers of Western Michigan PC, Grand Rapids, Michigan
  - Henry Ford Providence Novi Hospital, Novi, Michigan
  - Henry Ford Providence Southfield CK Potluri Cancer Center, Southfield, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Astera Cancer Care, East Brunswick, New Jersey
  - Christus St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - NYU Langone Hospital Long Island, Mineola, New York
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Durham VAMC, Durham, North Carolina
  - Novant Health Zimmer Cancer Institute, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - OhioHealth, Columbus, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Joe Arrington Cancer Research Treatment Center, Lubbock, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Alexander T. Augusta Military Medical Center, Fort Belvoir, Virginia
  - Virginia Oncology Associates Brock Cancer Center, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown
  - Barwon Health - University Hospital Geelong, Geelong
  - Liverpool Hospital, Liverpool
  - Sir Charles Gairdner Hospital, Nedlands
  - Calvary Mater Newcastle Hospital, New South Wales
  - Wollongong Hospital, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Austria (4):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - SCRI CCCIT gem GmbH, Salzburg
  - Medical University Vienna, Vienna
  - Hanusch Krankenhaus, Vienna
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - ZAS Cadix, Antwerp
  - Ghent University Hospital, Ghent
  - Jolimont, Haine Saint Paul La Louviere
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - GZA Ziekenhuizen- Campus St Augustinus, Wilrijk
- Brazil (12):
  - Fundacao Pio XII, Barretos
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Instituto Do Cancer Do Ceara, Fortaleza
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Complexo Hospitalar de Niteroi, Niterói
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Hospital Sao Rafael, Salvador
  - Hospital Nove de Julho, São Paulo
  - Clinica Medica Sao Germano S/S LTDA, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CHU de Quebec L Hotel Dieu de Quebec, Québec, Quebec
- China (32):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Tongren Hospital CMU, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South Hospital, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - Beijing Chaoyang Hospital, Chaoyang District
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Meidical University Union Hospital, Fuzhou
  - Nanfang Hospital, Guangzhou
  - Sun Yat -Sen University Cancer Center, Guangzhou
  - No.1 Affiliated Hospital, Medical College of Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Qilu Hospital of Shandong University, Jinan
  - The First Affliated Hospital Of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Fourth People s Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Tongji Hospital Tongji Medical College, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The first affiliated hospital of xiamen university, Xiamen
  - Henan Cancer Hospital, Zhengzhou
- Czechia (6):
  - Fakultni nemocnice Brno, Brno-Bohunice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Pilsen
  - VFN v Praze, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Regionshospitalet Godstrup, Herning
  - Zealand University Hospital, Roskilde
  - Vejle Sygehus, Vejle
- France (10):
  - CHU Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - CHU Nantes, Nantes
  - CHU Hopital Saint Antoine, Paris
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - CHU de Rennes - Hopital Pontchaillou, Rennes
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
- Germany (7):
  - Helios Kliniken Berlin Buch Gmbh, Berlin
  - Med. Universitatsklinik Essen, Essen
  - Universitaetsklinikum Halle Saale, Halle
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg
  - Klinikum Nuernberg Nord, Nuremberg
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - Alexandra General Hospital of Athens, Athens Attica
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - G Papanikolaou Hospital of Thessaloniki, Thessalonikis
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - A O U Sant Orsola Malpighi, Bologna
  - Careggi University Hospital, Florence
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera di Rilievo Nazionale A Cardarelli, Naples
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Universita Degli Studi di Roma Tor Vergata, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Japan (21):
  - Juntendo University Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Kameda Medical Center, Chiba
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Kansai Medical University Hospital, Hirakata
  - Hyogo Medical University Hospital, Hyôgo
  - Saitama Medical University Hospital, Iruma-gun
  - Tokai University Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - Kumamoto University Hospital, Kumamoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - National Hospital Organization Shibukawa Medical Center, Shibukawa
  - Japanese Red Cross Medical Center, Shibuya-ku
  - Shizuoka Cancer Center, Sunto Gun
  - Fujita Health University Hospital, Toyoake
  - Yamagata University Hospital, Yamagata
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Netherlands (5):
  - VUMC Amsterdam, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Reinier de Graaf Gasthuis, Delft
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Zuyderland Medical Center, Sittard-Geleen
- Norway (2):
  - Oslo University Hospital HF Ulleval sykehus, Oslo
  - St. Olavs Hospital, Trondheim
- Poland (11):
  - Wojewodzki Szpital Kliniczny w Bialej Podlaskiej, Biała Podlaska
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Szpital Uniwersytecki nr 2 im. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne, Warsaw
  - Szpital Uniwersytecki im Karola Marcinkowskiego w Zielonej Gorze, Zielona Góra
- Portugal (4):
  - Uls Braga - Hosp. Braga, Braga
  - Champalimaud Foundation Champalimaud Centre, Lisbon
  - Instituto Portugues de Oncologia, Porto
  - Uls Hosp Sao Joao, Porto
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (14):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Institut Catala d Oncologia L Hospitalet, Barcelona
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Clinico Univ. de Valencia, Valencia
- Sweden (4):
  - Falu Lasarett, Falun
  - Skanes universitetssjukhus, Lund
  - Universitetssjukhuset Orebro, Örebro
  - Karolinska University Hospital Huddinge, Stockholm
- Switzerland (2):
  - Inselspital Universitatsspital Bern, Bern
  - Kantonsspital St Gallen, Sankt Gallen
- Turkey (Türkiye) (8):
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Liv Hospital Ankara, Ankara
  - Memorial Antalya Hospital, Antalya
  - Pamukkale University Medical Faculty, Denizli
  - Medipol University Hospital, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Ondokuz Mayis University, Samsun
- United Kingdom (9):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - University Hospitals Bristol and Weston, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Western General Hospital, Edinburgh
  - University College London Hospitals, London
  - Imperial College Healthcare, London
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency